CLINICAL TRIAL: NCT06726798
Title: Prospective Cohort Study on the Safety and Efficacy of Endorobotics for Endoscopic Submucosal Dissection (Endorobotics ESD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Dean, Faculty of Medicine, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUHK EndoRobotics
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Endoscopic submucosal dissection
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic ESD arm (Experimental)
  Interventions: Procedure: Endoscopic submucosal dissection with EndoRobotics traction device

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection with EndoRobotics traction device — All patients received robotic ESD under general anesthesia or monitored anaesthetic care at the endoscopy center of Prince of Wales Hospital. The targeted lesion would first be localized and pre-injected using a mixture of normal saline, indigocarmine, epinephrine and sodium hyaluronate. The robotic endoscopic traction device was then inserted to reach the target. Mucosal incision first started from the anal side followed by lifting with the grasper[Figure 1; Video 1]. Vio 3 diathermy system (ERBE, Germany) was used with endocut Q effect 3 and forced coagulation effect 3. Further submucosal dissection would be performed by electrocautery knife with traction achieved via EndoRobotics traction. Upon completion, the specimen would be retrieved upon withdrawal of the whole system.

SUMMARY:
This trial is a prospective, single arm study of 30 patients recruited to undergo endoscopic submucosal dissection (ESD) with a novel robotic assisted technology. It will assess the safety and performance of robotic-assisted endoscopic submucosal dissection (ESD) of superficial gastric and colorectal lesions that otherwise cannot be optimally and radically removed by snare-based techniques. The primary outcome of the study is rate of complete (R0) resection of the neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endoscopic diagnosis of early gastric or colorectal neoplasia
* Patients will be recruited according to ESGE and JGES guidelines for gastric & colorectal ESD including: 1. Lesions for which en bloc resection with snare EMR is difficult to apply; 2. Mucosal tumors with submucosal fibrosis; 3. Sporadic tumors in conditions of chronic inflammation and 4. Local residual or recurrent early carcinomas after endoscopic resection.

Exclusion Criteria:

* Informed consent not available
* Carcinoma of colon or rectum or stomach with invasion to submucosa or beyond
* Evidence of distant metastasis
* Presence of another active malignancy
* Pregnancy
* Patients unfit for general anesthesia
* Endoscopic platform cannot reach target lesion
* Patients recruited into another clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 30 days
  Rate of complete en bloc, one-piece resection with histologically-confirmed tumour-free lateral and vertical margins

SECONDARY OUTCOMES:
Rate of procedural haemorrhage | 30 days
  Hemorrhage at the resection site that requires transfusion, discontinuation of the procedure, or adjunctive open surgical control of haemorrhage, subcategorized by: Bleeding during the index procedure, or bleeding that occurs after the subject has left the procedure room after the index procedure.
Rate of adjunctive procedure requirement | 30 days
  Need of adjunctive procedures, during study procedure required to control bleeding (e.g. clips or haemostatic agents)
All cause mortality rate | up to 5 years
  Mortality rate after procedure
Rate of infection | up to 12 months
  Clinical sepsis with changes in inflammatory markers (WCC, CRP, temperature)
Duration of procedure | 1 day
  Total time of ESD procedure
Length of hospital stay | 3 months
  Length of hospital stay (in days)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided